CLINICAL TRIAL: NCT06917625
Title: Long Term Neurodevelopmental Impact of the Type of Feeding During the First Year of Life Neuroimaging and Electrophysiology Follow up Study
Brief Title: Follow up of Long Term Neurodevelopmental Impact of the Type of Feeding During the First Year of Life at 10 Years Old
Status: Active, not recruiting | Type: Observational
Sponsor: Corporación de Apoyo de la Investigación Científica en Nutrición (Other)
Responsible Party: Principal Investigator, Cecilia Algarin, Adjunct Professor, Corporación de Apoyo de la Investigación Científica en Nutrición
Other Study IDs: MJCINUT8736
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Child Development
Keywords: early nutrition; brain development
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FM EM: During the first year of life the participants received
  1. regular formula milk
  2. enriched with Milk Fat Membrane Globule formula
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — The participants will be assessed with a brain MRI and will performed a neurophysiological test to evaluate executive functions
  Other Names: Event related potential test

SUMMARY:
The Chilean infant Nutrition Trial was a prospective, randomized, double-blind, controlled study conducted in Santiago, Chile, between 2016 and The study aimed to evaluate growth and body composition changes between birth and two years of age in a large sample of children who were randomized to receive either infant formula with or without added MFGM (milk fat globule membrane) through 12 months of age or received human milk as part of the reference group. In a subsample of 160 children, neurodevelopmental were assessed at 6 months and 24 months.

DETAILED DESCRIPTION:
To test our hypothesis, this study proposes to investigate our conceptual model's direct and indirect associations using a combination of low-field MRI, electrophysiology, and psychometric assessments of executive functioning and general cognitive development, expecting to re-enroll approx 100 participants. These children will undergo ERPs, low-field MRI and neurocognitive testing to evaluate brain structure, function, and cognitive development.

The Go/No-Go task assesses inhibitory control, one of the most important executive function. Its development has been studied electrophysiologically using event-related potentials (ERPs), in tasks that require active inhibition when there is a previously learned or prepotent response. The main relevant ERP components are the N2 and P300. The N2, an early negative deflection, has been interpreted to reflect attention, the P300, a later positive wave, is thought to reflect resource allocation. The P300 is typically greater in the inhibitory than in the prepotent response components of tasks such as the Go/No-Go task. Behavioral responses such as accuracy and reaction time have also been studied as measures of development (2). Using the collected data, inhibitory control, as one of the earliest executive functions to begin developing, will be studied.

The data acquired with the Low-field MRI quantify and compare brain structure and myelination patterns (derived from MRI) across the feeding groups in specific white matter pathways and brain regions involved in executive function (EF) and throughout the brain generally. MRI comparisons and comparisons will be complemented by comparisons of ERP measures collected during an inhibition task, which assesses functional development and processing speed.In addition to these group-wise comparisons,it will be explored the direct and indirect infant feeding -> brain structure and function -> executive function and cognitive performance associations using a series of ANCOVA and general linear modeling methods.

C. PRIMARY OBJECTIVE AND OUTCOME MEASUREMENTS:

The primary objective of this study is to determine whether additional intake of bMFGM during infancy (0-12 months of age) improves brain structure, function, and cognitive performance (specifically EF) at early school age (8-10 years of age).

The following measures will be collected, and EF domains assessed and comparisons made.

Brain Structure and Myelin Imaging. Low-Field MRI will be used to assess general brain growth and morphometry (total brain volume, whole-brain white and gray matter volume, and cortical and sub-cortical structure volumes) as well as myelination using myelin-sensitive MRI. Differences across all of these measures between the infant feeding groups (standard formula, added bMFGM, and breastfeeding reference) will be part of exploratory analysis. To examine specific hypothesized brain regions involved in EF, including prefrontal cortex, hippocampus, amygdala, thalamus, motor and somatosensory cortices, and auditory cortex will be studied. Connecting white matter regions, including corpus callosum, cingulum, superior longitudinal fasciculus, and anterior thalamic radiations will be compared as they are an indirect index of myelination grade.

Mean myelin measures will be calculated for each white matter pathway and compared across the three feeding groups using an ANCOVA and post hoc Tukey test to identify significant differences.

ERPs and Electrophysiology. ERPs will be recorded from 128 scalp sites using a recording system with a geodesic sensor net (Electric Geodesic, Inc., Eugene, Oregon). The vertex was used as the on-line reference electrode. The signal was sampled at 1000 Hz and bandpass filtered at 0.1 to 100 Hz. After recording, stimulus triggers were exported and analyzed using signal processing software (BESA Research 6.1 BESA® ,Germany). Signals were re-referenced off-line to an average (whole head) reference and bandpass filtered (0.1 to 10 Hz). The continuous EEG was segmented into epochs according to the three stimulus types: block 1 Go trials, block 2 Go trials, and block 2 No-Go trials with the segment length being the same as each onset-to-onset interval. Noisy segments of data with excessive electromyographic signal (EMG) were rejected by visual inspection, and noisy channels were identified and rejected using a 2.5% probability threshold and visual inspection. Each trial will last 1000ms and consist of 100ms of pre-stimulus presentation, 500ms of stimulus presentation, and 1000ms of stimulus recording. The intertrial interval was 500 to 700ms. For the ERP analysis, window time was selected to establish where to determine the components of interest, which were identified relative to the number of major positive and negative peaks following stimulus onset. All time window values were relative to stimulus onset, and the peak amplitudes were calculated relative to the baseline amplitude. Statistical analyses were conducted with SPSS software version 25.0.1 (SPSS Inc., Chicago, IL, USA). Behavioral measures were reaction time and accuracy. Electrophysiological measures were peak amplitude and latency for N2 and amplitude for P300. Covariates that indicated group differences were considered in subsequent analyses as potential confounders.

Age-appropriate EF Psychometric Assessments will be used to evaluate executive functions. The EFECO assessment that are the abbreviation Evaluation of executive function throughout conductual observation. The questionnaire will be filled by the adult in charge of the participant.

ELIGIBILITY:
Inclusion Criteria: Healthy, have been studied at 2 and 6 years old in the laboratory -

Exclusion Criteria: To have a diagnosis of a neurological disease.

-

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population was selected from the neighborhoods close to the installation of research institute. The area corresponds to the southeast of Santiago, Chile
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To determine if intake of bMFGM during the first year improves brain structure at 9 ys. | MRI assessment will be performed at 9 years old in a session of 45 minutes
  Low-Field MRI will be used to assess general brain growth and morphometry (total brain volume, whole-brain white and gray matter volume, and cortical and sub-cortical structure volumes) as well as myelination using myelin-sensitive MRI. For specific analysis will examine brain regions involved in EF, including prefrontal cortex, hippocampus, amygdala, thalamus, motor and somatosensory cortices, and auditory cortex ; and connecting white matter regions, including corpus callosum, cingulum, superior longitudinal fasciculus, and anterior thalamic radiations .The results will be expressed by mean volumetric measures calculate from the MRI data using validated FreeSurfer software and compared across the groups using an ANCOVA, controlling for variables of interest. Mean myelin measures will be calculated for each white matter pathway and to identify significant differences (express by grade of myelination)
To determine if intake of bMFGM during the first year improves EF measures by ERPs at 9ys. | ERPs assessment will be performed at 9 years old in a a second session of 90 minutes .
  . To assess EF the Go No Go task will be performed with ERPs. The participant will ask to press a button when any letter appears (Go stimulus) except when the letter will be X (No Go stimulus). There will be 2 blocks: Block 1(40 trials) of Go stimulus and Block 2 (200 trials) of randomized Go and No Go stimuli. Neurophysiological responses will be recorded from 128 scalp sites using a recording system with a geodesic sensor net .For the ERP analysis, the major positive and negative peaks following stimulus onset will be identified. Statistical analyses were conducted with SPSS software version 25.0.1. Behavioral measures will be reaction time (ms) and accuracy (%). Electrophysiological results will be the peak amplitude (mµ) and latency (ms) for the waves N2 and P300.
To determine if intake of bMFGM during the first year improves EF measures by questionnaire EFECO. | EFECO will be answered by the adult that ERPs assessment will be performed at 9 years old in a a second session of 90 minutes .
  The questionnaire EFECO evaluates executive functions throughout conductual observation.
  The scale has 67 questions which measure seven different executive functions: cognitive flexibility, emotional control, planification capacity, organization, initiative and working memory. The quantification of each item goes from 0 to 3 according with one of these responses: Never, sometime, frequently, and very frequently. The higher score corresponds to a better EF. The questionnaire will be filled by the adult accompanying the participant during the ERP measurement and confirm that lives with the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Peirano, MD, Study Director — University of Chile
Locations (1):
- CINUT, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
The data published in an article could be share with other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and 1 year after the publication
Access Criteria: By a written request to the authors